CLINICAL TRIAL: NCT04641130
Title: Validation and Reproducibility Study of the ALYATEC Allergen Exposure Chamber by Determining the Concentration of Birch Pollen Allergen Inducing Conjunctivitis in Subjects Allergic to Birch Pollen.
Brief Title: Clinical Validation Study in Allergic Conjunctivitis to Birch Pollen During Allergen Challenge in ALYATEC EEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alyatec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ALY-002B
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Allergic Conjunctivitis
Keywords: Allergy; Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic; Hypersensitivity; Conjunctivitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposure to birch pollen (Experimental): Step 1: dose validation 16 subjects are exposed for 2 consecutive days (D1 + D2), to the same aerial concentration of Bet v1.
  The main objective is achieved if the Abelson score is ≥ 5 on J1 or J2. If the main objective is achieved for the 60 ng/m3 concentration, 8 responder subjects will directly perform step 2.
  If the main objective is not achieved for the 60 ng/m3 concentration, the subjects will be exposed between 7 to 10 days after exposure 1, to an allergen concentration of 120 ng/m3 (Exposure 2: D1 + D2).
  Step 2: reproducibility Once the allergen concentration has been determined (step 1), 8 of the responder subjects from step 1 are exposed again to this same concentration, during 2 additional exposures (Exposure 3: D1 + D2 and Exposure 4: D1 + D2), at least 7 days apart.
  A wash-out period of at least 7 days is observed between step 1 and 2. The duration of allergen exposure will be a maximum of 4 hours for all exposures.
  Interventions: Other: Exposure to birch pollen in EEC

INTERVENTIONS:
Other: Exposure to birch pollen in EEC — Patients are exposed to airborne birch pollen allergen. The duration of each exposure is 4h maximum.

SUMMARY:
This is a single center open study designed to determine the concentration of airborne birch pollen inducing an allergic conjunctivitis response in individuals allergic to birch pollen, during allergen exposures in the Alyatec environmental exposure chamber (EEC).

ELIGIBILITY:
Inclusion Criteria:

* Subjects having signed the informed consent
* Subjects affiliated to a social security scheme
* Subjects with birch pollen rhinitis and conjunctivitis with:
* A history of rhinoconjunctivitis for at least the last 2 consecutive pollen seasons.
* A positive skin prick-test to birch (wheal diameter >6 mm compared to the negative control),
* Specific immunoglobulin E (IgE) for birch> 0.1 kIU/l
* Women of childbearing potential must have a negative pregnancy test during the entire study period with an effective means of contraception: oral contraceptives, intrauterine device, condom with spermicide for at least one month before inclusion in the study and for the duration of the study. At each study visit and each exposure on D1, a urine pregnancy test will be performed.
* A positive conjunctival provocation test to birch during the screening visit at a dilution of 100IR/ml maximum

Exclusion Criteria:

* Known asthmatic subjects allergic to birch pollen
* Use of oral corticosteroids in the 4 weeks preceding inclusion in the study
* Use of biotherapy in the 4 months preceding inclusion in the study
* Desensitization to birch pollen in the last 5 years
* Uncontrolled chronic pathologies (hypertension, cardiac, respiratory, renal pathology).
* Active autoimmune disease
* Uncontrolled systemic hypertension
* Subjects who participated in another clinical study in the three months prior to inclusion
* Pregnancy and breast feeding
* Inability to understand and act upon the information provided

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Determine the concentration of birch pollen allergen (in ng/m3 of Bet v1) necessary to induce a conjunctival response in at least 50% of subjects allergic to birch. | 4 hours exposure in EEC
  A positive conjunctival response is defined by an Abelson score ≥ 5.

SECONDARY OUTCOMES:
Evaluate the reproducibility of allergen exposure in the ALYATEC EEC | 4 hours exposure in EEC
  The reproducibility of the exposure will be assessed by measuring the quantity of birch pollen allergen (ng Bet v1) inducing a conjunctival response during step 2.
Study the effect of EEC birch pollen exposure on symptoms of rhino-conjunctivitis. | 4 hours exposure in EEC
  The effect of the exposure on the rhinoconjunctival response will be assessed by Rhinoconjunctivitis Total Symptom Score (RTSS).
  The RTSS is the sum of 6 rhinoconjunctivitis symptom scores: sneezing, rhinorrhea, nasal pruritus, nasal congestion, ocular pruritus and watery eyes.
  Each symptom is graded in a 4-point scale as follows: 0: no symptoms, 1: mild symptoms, 2: moderate symptoms, 3: severe symptoms. It ranges from 0 to 18. The lower the score, the better the outcome.
Study the effect of EEC birch pollen exposure on symptoms of rhinitis | 4 hours exposure in EEC
  The effect of the exposure on the rhinitis response will be assessed by rhinitis Visual Analogue Scale (VAS).
  The rhinitis VAS is a measurement of patient's subjective evaluation of symptoms severity. Patients will score the severity of their nasal symptoms on a scale, with 0 meaning no symptoms and 10 meaning the worst symptoms.
Study the effect of EEC birch pollen exposure on symptoms of conjunctivitis. | 4 hours exposure in EEC
  The effect of the exposure on the conjunctival response will be assessed by Conjunctivitis Visual Analogue Scale (VAS).
  The conjunctivitis VAS is a measurement of patient's subjective evaluation of symptoms severity. Patients will score the severity of their ocular symptoms on a scale, with 0 meaning no symptoms and 10 meaning the worst symptoms.
Measure the amount of particles carrying the allergens. | 4 hours exposure in EEC
  The amount of particles carrying the allergen will be measured with counters located in the exposure chamber.
Measure the aerodynamic diameter of the particles carrying the allergens. | 4 hours exposure in EEC
  The aerodynamic diameter of the particles carrying the allergen will be measured with counters located in the exposure chamber.
Evaluate changes in mitochondrial respiration | 4 hours exposure in EEC
  The changes in mitochondrial respiration will be done by evaluating the modifications of the I to IV complex of the mitochondrial respiratory chain, before and after allergen exposure

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric de Blay, Pr., Principal Investigator — Alyatec
Locations (1):
- Alyatec, Strasbourg, Grand Est, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alyatec website — https://www.alyatec.com/en/